CLINICAL TRIAL: NCT00973817
Title: Efficacy and Safety of the Extracorporeal Liver Assist Device (ELAD) in Subjects With Acute On Chronic Hepatitis (AOCH)
Brief Title: Efficacy and Safety of the Extracorporeal Liver Assist Device (ELAD) in Acute on Chronic Hepatitis
Acronym: SILVER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vital Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTI-206
Record Dates: First submitted 2009-09-02; First posted 2009-09-09 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Acute On Chronic Hepatitis
Keywords: Hepatitis; AOCH
MeSH Terms: conditions — Hepatitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELAD (Experimental): Use of ELAD for up to 6 days to stabilize liver function plus standard of care treatment plus standard of care treatment. Standard of care for acute on chronic hepatitis patients including medications and treatments typically given to patients admitted with acute hepatitis (Pentoxifylline, corticosteroids, abdominal paracentesis, nutritional therapy, etc., if indicated)
  Interventions: Biological: ELAD plus standard of care treatment; Other: Standard of care
- Standard of care (Other): Standard of care for acute on chronic hepatitis patients including medications and treatments typically given to patients admitted with acute hepatitis (Pentoxifylline, corticosteroids, abdominal paracentesis, nutritional therapy, etc., if indicated)
  Interventions: Other: Standard of care

INTERVENTIONS:
Biological: ELAD plus standard of care treatment — Use of ELAD plus standard of care
  Other Names: Extra corporeal liver assist system
  Arms: ELAD
Other: Standard of care — Standard of care in the treatment of AOCH will be administered

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of the use of ELAD in patients with diagnosed Acute On Chronic Hepatitis, including Acute Alcoholic Hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18</= 67 years; AND
* Acute decompensation of chronic liver disease over the preceding 30 days; AND
* MELD score between 18 and 35, inclusive; AND
* Subject or designated representative must provide Informed Consent

Exclusion Criteria:

* Platelets <50,000mm at baseline; OR
* Evidence of chronic renal failure as defined by a serum creatinine >/= 2.5mg/dL as measured during the 1-6 month period prior to study entry. (Subject is not excluded with a creatinine >2.5 mg/dL if deemed to be type-1 hepato-renal syndrome); OR
* Contraindication to renal replacement therapy (hemodialysis or hemofiltration); OR
* International Normalization Ratio (INR) > 3.5; OR
* Septic shock as defined by a positive blood culture and two or more of the following:

  * Systolic blood pressure <90mmHg OR mean arterial pressure <60mmHg;
  * Tachypnea > 20 breaths per minute OR a PaCO2<32 mmHg;
  * White blood cell count < 4000 cell/mm3 OR > 12000 cell/mm3 (<4 x 10(9) or >12 x 10(9) cells/L).
* Evidence of major hemorrhage as indicated by:

  * requiring >/= 4 units packed red blood cells within a 48 hour period prior to Screening, OR
  * hemodynamic instability (sustained pulse > 120 beats/min AND systolic blood pressure < 100 mmHg over one hour)

Subjects with a recent history of gastrointestinal hemorrhage who have been successfully treated and remain hemodynamically stable for a period of 48 hours will then be eligible for the study if the investigator determines the subject to be at low risk for rebleeding; OR

* Evidence (by physical exam, history or lab evaluation) of significant concomitant disease including chronic congestive heart failure, vascular disease, emphysema, AIDS, hepatitis due to herpes virus, Wilson's disease, or Budd-Chiari syndrome; OR
* Known history of hepatocellular carcinoma beyond the Milan criteria and/or portal vein thrombosis; OR
* Evidence of spontaneous bacterial peritonitis with uncontrolled infection; OR
* Evidence of brain death as determined by blood flow studies positive for herniation AND/OR absence of pupillary reflex; OR
* Systolic blood pressure <85 mmHg OR MAP <50mmHg at baseline; OR
* Requirement for escalating doses of vasopressor support OR of an alpha-adrenergic agent for one hour or longer AND evidence of hemodynamic instability; OR
* Subject at maximum vasopressor dose at Screen; OR
* Clinical or radiographic evidence of a new stroke or intracerebral bleeding; OR
* Seizures uncontrolled by medication; OR
* Acute myocardial infarction based on clinical and/or electrocardiographic evidence; OR
* Lung disease defined by a PaO2<60mmHg on room air, acute respiratory distress syndrome, or a history of severe COPD or interstitial lung disease; OR
* Pregnancy as determined by beta-HCG results or lactation; OR
* Participation in another investigational drug, biologic, or device study within 1 month of enrollment. Subjects enrolled in an observational study will be eligible for this trial.
* Previous liver transplant.
* Previous participation in a clinical trial involving ELAD.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Time to progression at which a 5-point or greater Model for End stage Liver Disease (MELD) score is recorded relative to baseline | From Baseline up to Study Day 91
  This is based on death or the first observed increase of at least 5 points from Baseline MELD score (whichever occurs earlier) at least 24 hours after the ELAD® Treatment Period is ended and up to Study Day 91 (90 days following Baseline).

SECONDARY OUTCOMES:
Time to progression at which a 5-point or greater MELD score is recorded relative to baseline | From Baseline up to Study Day 91
  A secondary Overall Survival analysis will use the same methodology as the primary time to progression efficacy analysis, except that an event will be defined as death. Secondary efficacy analyses will evaluate the proportion of progression free survivors (MELD score increased less than 5 points relative to the Baseline MELD score).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ashley, MS, Study Director — Vital Therapies, Inc.
Locations (21):
- United States (15):
  - Cedars Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - New York University Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Univ. of Rochester, Strong Memorial Hospital, Rochester, New York
  - Westchester Medical Center, Valhalla, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
- United Kingdom (6):
  - University Hospitals Birmingham, Birmingham, England
  - Kings College Hospital NHS Foundation Trust, London, England
  - Royal Derby Hospital, Derby
  - Edinburgh Royal Infirmary, Edinburgh
  - St. James University Hospital, Leeds
  - Royal Free Hospital London, London